CLINICAL TRIAL: NCT01064856
Title: A Multicenter Study of the Efficacy and Safety of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Peripheral Spondyloarthritis
Brief Title: Study of Adalimumab in Participants With Peripheral Spondyloarthritis (SpA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-883; 2009-014567-39 (EudraCT Number)
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Spondyloarthritis
Keywords: peripheral spondyloarthritis; adalimumab; humira
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Double-blind (DB) Adalimumab (Experimental): Adalimumab 40 mg subcutaneous (SC) injection every other week (eow) up to Week 12 in double-blind period.
  Interventions: Biological: Adalimumab
- Double-blind Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection every other week (eow) up to Week 12 in the double-blind period.
  Interventions: Biological: Placebo
- Double-blind Adalimumab / Open-label Adalimumab (Experimental): Adalimumab 40 mg SC injection eow up to Week 12 in double-blind period and from Week 12 to Week 156 in open-label period.
  Interventions: Biological: Adalimumab
- Double-blind Placebo / Open-label Adalimumab (Placebo Comparator): Placebo SC injection every other week (eow) up to Week 12 in the double-blind period; adalimumab 40 mg subcutaneous injection eow from Week 12 to Week 156 in the open-label period.
  Interventions: Biological: Adalimumab; Biological: Placebo

INTERVENTIONS:
Biological: Adalimumab — Study drug was provided as a sterile SC injection solution in 1 mL pre-filled syringes containing adalimumab 40 mg/0.8 mL. Study drug was SC self-administered eow at approximately the same time of day.
  Other Names: ABT-D2E7; Humira
  Arms: Double-blind (DB) Adalimumab; Double-blind Adalimumab / Open-label Adalimumab; Double-blind Placebo / Open-label Adalimumab
Biological: Placebo — Study drug was provided as a sterile SC injection solution in 1 mL pre-filled syringes containing matching placebo for adalimumab. Study drug was SC self-administered eow at approximately the same time of day.
  Arms: Double-blind Placebo; Double-blind Placebo / Open-label Adalimumab

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of adalimumab 40 mg administered every other week (eow) subcutaneously (SC) compared to placebo for 12 weeks followed by open label (OL) safety and efficacy assessments in participants with non-ankylosing spondylitis (AS), non-psoriatic arthritis (PsA) active peripheral spondyloarthritis (SpA) who have had an inadequate response to >= 2 non-steroidal anti-inflammatory drugs (NSAIDs), or are intolerant to, or have a contraindication for, NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants who had inadequate response to >= 2 non-steroidal anti-inflammatories (NSAIDs)
* Participants who had arthritis or enthesitis or dactylitis plus: met spondyloarthritis clinical criteria
* Negative purified protein derivative (PPD) test and Chest X-Ray performed at Baseline Visit were Negative
* Ability to administer subcutaneous injections
* General good health

Exclusion Criteria:

* Prior anti-tumor necrosis factor (TNF) therapy
* Psoriasis or Psoriatic Arthritis
* Fulfillment of modified New York criteria for Ankylosing Spondylitis
* Recent infection requiring treatment
* Significant medical events or conditions that had put patients at risk for participation
* Female participants who were pregnant or breast-feeding or considering becoming pregnant during the study
* History of cancer, except successfully treated skin cancer
* Recent history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In-Ho Song, MD, Study Director — AbbVie

REFERENCES:
- [Background] Mease P, Sieper J, Van den Bosch F, Rahman P, Karunaratne PM, Pangan AL. Randomized controlled trial of adalimumab in patients with nonpsoriatic peripheral spondyloarthritis. Arthritis Rheumatol. 2015 Apr;67(4):914-23. doi: 10.1002/art.39008. PMID 25545240
- [Derived] Coates LC, Abraham S, Tillett W, Mease PJ, Ramiro S, Wu T, Wang X, Pangan AL, Song IH. Performance and Predictors of Minimal Disease Activity Response in Patients With Peripheral Spondyloarthritis Treated With Adalimumab. Arthritis Care Res (Hoboken). 2022 Feb;74(2):259-267. doi: 10.1002/acr.24442. Epub 2021 Dec 29. PMID 32937016
- [Derived] Mease PJ, Van den Bosch F, Sieper J, Xia Y, Pangan AL, Song IH. Performance of 3 Enthesitis Indices in Patients with Peripheral Spondyloarthritis During Treatment with Adalimumab. J Rheumatol. 2017 May;44(5):599-608. doi: 10.3899/jrheum.160387. Epub 2017 Mar 15. PMID 28298558
- [Derived] Turina MC, Ramiro S, Baeten DL, Mease P, Paramarta JE, Song IH, Pangan AL, Landewe R. A psychometric analysis of outcome measures in peripheral spondyloarthritis. Ann Rheum Dis. 2016 Jul;75(7):1302-7. doi: 10.1136/annrheumdis-2014-207235. Epub 2015 Aug 5. PMID 26245756
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Double-blind (DB) Period
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo | Double-blind Adalimumab / Open-label Adalimumab | Double-blind Placebo / Open-label Adalimumab
Started | 84 | 81 | 0 (This treatment group is not applicable for this period.) | 0 (This treatment group is not applicable for this period.)
Completed | 82 | 81 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Consent withdrawn by participant | 1 | 0 | 0 | 0
Period: Open-label (OL) Period
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo | Double-blind Adalimumab / Open-label Adalimumab | Double-blind Placebo / Open-label Adalimumab
Started | 0 (This treatment group is not applicable for this period.) | 0 (This treatment group is not applicable for this period.) | 82 | 81
Completed | 0 | 0 | 56 | 61
Not Completed | 0 | 0 | 26 | 20
Not completed — Adverse Event | 0 | 0 | 12 | 6
Not completed — Consent withdrawn by participant | 0 | 0 | 5 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug (ITT).
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo | Total
Number analyzed (Participants) | 84 | 81 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.79) | 38.5 (12.77) | 40.6 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 36 | 39 | 75
Tender Joint Count (78 Joints) [Mean (Standard Deviation); unit: units on a scale] — Seventy-eight joints were assessed for tenderness by physical examination. Tenderness of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with tenderness) to 78 (worst possible score/ 78 joints with tenderness).
  units on a scale | 12.95 (12.79) | 13.62 (16.10) | 13.28 (14.46)
Swollen Joint Count (76 Joints) [Mean (Standard Deviation); unit: units on a scale] — Seventy-six joints were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with swelling) to 76 (worst possible score/ 76 joints with swelling).
  units on a scale | 6.12 (5.58) | 7.31 (7.99) | 6.70 (6.87)
Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) [Mean (Standard Deviation); unit: units on a scale] — Assessment of enthesitis was performed in 7 domains. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total MASES ranging from 0 (0 sites with tenderness) to 13 (worst possible score; 13 sites with tenderness).
  units on a scale | 3.13 (3.60) | 3.59 (3.39) | 3.36 (3.50)
Leeds Enthesitis Index [Mean (Standard Deviation); unit: units on a scale] — Assessment of enthesitis was performed in 6 domains. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total Leeds Enthesitis Index scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
  units on a scale | 1.49 (1.66) | 1.42 (1.61) | 1.45 (1.63)
Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Score [Mean (Standard Deviation); unit: units on a scale] — Assessment of enthesitis was performed in 16 domains. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total SPARCC scores ranging from 0 (0 sites with tenderness) to 16 (worst possible score; 16 sites with tenderness).
  units on a scale | 3.83 (4.03) | 4.05 (3.78) | 3.94 (3.90)
Total Enthesitis Count [Mean (Standard Deviation); unit: units on a scale] — Total enthesitis count in the sum of all unique, individual enthesis location included in the Leeds, SPARCC and MASES entheses indices. Scores range from 0 (0 sites with enthesitis) to 29 (29 sites with enthesitis).
  units on a scale | 6.73 (6.95) | 7.33 (6.69) | 7.02 (6.81)
Patient Global Assessment (PTGA) of Disease Activity [Mean (Standard Deviation); unit: mm] — PTGA of Disease Activity as measured by a 100 mm visual analogue scale (VAS) where 0=no symptoms and 100=maximum symptoms.
  mm | 65.24 (15.22) | 66.43 (15.86) | 65.82 (15.50)
PTGA - Pain [Mean (Standard Deviation); unit: units on a scale] — PTGA - Pain as measured by a 100 mm VAS where 0=no pain and 100=maximum pain.
  units on a scale | 64.30 (14.03) | 65.60 (15.89) | 64.94 (14.94)
Physician Global Assessment (PGA) of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — PGA of Disease Activity as measured by a 100 mm VAS where 0=no symptoms and 100=maximum symptoms.
  units on a scale | 60.29 (15.53) | 57.02 (14.98) | 58.68 (15.31)
Ankylosing Spondylitis Disease Activity Score (ASDAS) [Mean (Standard Deviation); unit: units on a scale] — The ASDAS is a continuous disease activity score: low score indicates lower disease activity and higher values indicate higher disease activity. The score ranges from 0 to no defined upper limit. It is categorized into 4 disease activity states based on score: inactive disease (< 1.3), moderate (≥ 1.3 to < 2.1), high (≥ 2.1 to ≤ 3.5), and very high (> 3.5). One participant in the Placebo arm did not have a baseline ASDAS assessment.
  units on a scale | 2.92 (0.84) | 3.06 (0.80) | 2.99 (0.82)
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Mean (Standard Deviation); unit: units on a scale] — The BASDAI consisted of a VAS scale used to answer 6 questions pertaining to symptoms experienced by the participant for the past week. Each question on the BASDAI was reported in centimeters (0 [none] to 10 [very severe] with one question's possible answers being in time increments [0 hours to ≥ 2 hours]). The overall BASDAI score ranges from 0 to 10 cm. Lower scores indicate less disease activity.
  units on a scale | 5.68 (1.74) | 5.57 (1.58) | 5.62 (1.66)
Dactylitis Count [Mean (Standard Deviation); unit: units on a scale] — Assessment of the presence or absence of dactylitis as well as grading of tenderness and swelling in all 20 of the participants' digits was performed. Tenderness at each site was quantified from absent to severe. Swelling was quantified from mild to severe. Total Dactylitis Assessment scores ranging from 0 (0 digits with dactylitis) to 20 (worst possible score; 20 digits with dactylitis). One participant in the Double-blind (DB) Adalimumab arm did not have a baseline dactylitis count.
  units on a scale | 0.35 (0.94) | 0.65 (1.25) | 0.50 (1.11)
Short Form-36 Health Status Survey™ Version 2 (SF-36™V2) Physical Component Score (PCS) [Mean (Standard Deviation); unit: units on a scale] — The SF-36™V2 is a 36-item generic health-related quality of life measure to assess the participant's view of their health consisting of 2 components: physical and mental. Scores range from 0 to 100. Higher scores indicate a better health state.
  units on a scale | 34.56 (7.93) | 34.48 (7.62) | 34.52 (7.76)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders According to the Composite Peripheral SpA Response Criteria (PSpARC 40) at Week 12
Description: Percentage of participants achieving the following composite response at Week 12: >= 40% improvement (minimum 20 mm absolute improvement) from Baseline in Patient Global Assessment (PTGA) of Disease Activity as measured by a 100 mm visual analogue scale (VAS) where 0=no symptoms and 100=maximum symptoms; >= 40% improvement (minimum 20 mm absolute improvement) from Baseline in PTGA - Pain as measured by a 100 mm VAS where 0=no pain and 100=maximum pain; and >= 40% improvement from Baseline in at least 1 of the following 3 criteria: swollen joint count (76 joints) and tender joint count (78 joints); total enthesitis count; or total dactylitis count. Non-responder imputation: missing response was imputed as non-response.
Time Frame: Week 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
percentage of participants
  Responder | 39.3 | 19.8
  Non-responder | 60.7 | 80.2
Statistical Analysis 1: Comparison: Double-blind (DB) Adalimumab vs Double-blind Placebo; Test type: Superiority or Other; p = 0.006, Pearson's chi-square

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with treatment. If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE): results in death or is life-threatening, results in admission or prolongation of hospitalization, results in congenital anomaly or persistent or significant disability/incapacity, or is an important medical event requiring medical or surgical intervention to prevent serious outcome. AEs were categorized by severity (mild, moderate, severe) and relationship to treatment (probably, possibly, probably not, not related). Please see Adverse Events section below for more details.
Time Frame: Baseline (day of first study drug administration) through Week 156 plus 70 days
Population: Safety Analyses included all participants who received at least 1 dose of double-blind study drug.
Measure: Number; unit: participants
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
participants
  Any adverse event | 47 | 45
  Any serious adverse event | 1 | 1
  Any AE leading to discontinuation of study drug | 3 | 0
  Any severe AE | 4 | 2
  Any AE at least possibly drug related | 21 | 15
  Any SAE at least possibly drug related | 0 | 0
  Any infection | 18 | 24

3. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) of Disease Activity at Week 12
Description: A VAS was to be used for the Physician Global Assessment (PGA) of disease activity (current status). The left end of the VAS scale (0 mm) signifies the absence of symptoms and the right end (100 mm) signifies maximum disease activity. Last observation carried forward (LOCF): missing values were imputed using the last non-missing post-baseline value prior to the missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -32.2 (22.52) | -18.2 (22.93)
Statistical Analysis 1: Comparison: Double-blind (DB) Adalimumab vs Double-blind Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; The P-value was based on an ANCOVA model adjusting for baseline with treatment as a factor

4. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 12
Description: The BASDAI was to be completed at the designated study visits. The participant was to assess his/her disease activity using the BASDAI which consisted of a VAS scale used to answer 6 questions (Q1 through Q6) pertaining to symptoms experienced by the participant for the past week. Each question on the BASDAI was reported in centimeters (0 [none] to 10 [very severe] with one question's possible answers being in time increments [0 hours to ≥ 2 hours]). The overall BASDAI score ranges from 0 to 10 cm and was calculated as follows: BASDAI Score = 0.2 × (Q1 + Q2 + Q3 + Q4 + Q5/2 + Q6/2). Lower scores indicate less disease activity. LOCF: Missing value was imputed using the last non-missing post-baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -2.1 (2.32) | -1 (2.19)
Statistical Analysis 1: Comparison: Double-blind (DB) Adalimumab vs Double-blind Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; The P-value was based on an ANCOVA model adjusting for baseline with treatment as a factor

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Modified for the Spondyloarthropathies (HAQ-S) Total at Week 12
Description: The HAQ-S is a self-reported measure to assess the physical function and health-related quality of life. The Disability Index (DI) of HAQ-S is calculated as the mean of the following 8 category scores (range: 0 [without any difficulty] to 3 [unable to do]): Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Five additional items in the functional status measure were included in the HAQ-S, including carrying heavy packages, sitting for long periods, able to work at a flat topped table, and (if the participant had a driver's license or a car) able to look in the rear view mirror and able to turn head to drive in reverse. The overall score ranges from 0 (no disability) to 3 (three very severe, high-dependency disability). Negative mean changes from Baseline in the overall score indicate improvement. LOCF: Missing value was imputed using the last non-missing post-baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -0.3 (0.44) | -0.2 (0.47)
Statistical Analysis 1: Comparison: Double-blind (DB) Adalimumab vs Double-blind Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA; The P-value was based on an ANCOVA model adjusting for baseline with treatment as a factor

6. Secondary Outcome: Change From Baseline in Short Form-36 Health Status Survey™ Version 2 (SF-36™V2) Physical Component Score (PCS) at Week 12
Description: The Short Form-36 Health Status Survey™ Version 2 (SF-36™V2) is a 36-item generic health-related quality of life measure to assess the participant's view of their health consisting of 2 components: physical and mental. For each component, a transformed summary score is calculated using 8 sub-domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100. Higher scores indicate a better health state.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug and had non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 83 | 79
units on a scale | 6.7 (7.85) | 2.4 (6.65)

7. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 12
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Each domain was graded for the presence (1) or absence (0) of tenderness yielding total MASES ranging from 0 (0 sites with tenderness) to 13 (worst possible score; 13 sites with tenderness). Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -1.2 (2.67) | -0.8 (2.38)

8. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index at Week 12
Description: Assessment of enthesitis was performed in the following 6 domains: left and right lateral epicondyle, left and right medial femoral condyle, left and right Achilles tendon insertion. Tenderness at each site was quantified on a dichotomous basis: Each domain was graded for the presence (1) and absence (0) of tenderness yielding total Leeds Enthesitis Index scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -0.8 (1.28) | -0.1 (1.19)

9. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Score at Week 12
Description: Assessment of enthesitis was performed in the following 16 domains: left and right (L/R) medial epicondyle; L/R lateral epicondyle; L/R supraspinatus insertion into the greater tuberosity of humerus; L/R greater trochanter; L/R quadriceps insertion into superior border of patella; L/R patellar ligament insertion into inferior pole of patella or tibial tubercle; L/R Achilles tendon insertion into calcaneum; L/R plantar fascia insertion into calcaneum. Tenderness at each site was quantified on a dichotomous basis. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total SPARCC scores ranging from 0 (0 sites with tenderness) to 16 (worst possible score; 16 sites with tenderness). Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -1.7 (2.43) | -0.7 (2.21)

10. Secondary Outcome: Change From Baseline in Dactylitis at Week 12
Description: Assessment of the presence or absence of dactylitis as well as grading of tenderness and swelling in all 20 of the participants' digits was performed. Tenderness at each site was quantified from absent to severe. Swelling was quantified from mild to severe. Total Dactylitis Assessment scores ranging from 0 (no digits with dactylitis) to 20 (worst possible score; 20 digits with dactylitis). Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug and had non-missing values for both Baseline and the post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 83 | 81
units on a scale | -0.2 (1.05) | 0.3 (0.93)

11. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 12
Description: Seventy-eight joints were assessed for tenderness by physical examination. Tenderness of each joint was classified as present (1) or absent (0), for a total possible TJC score of 0 (0 joints with tenderness) to 78 (worst possible score/78 joints with tenderness). Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 81
units on a scale | -5.9 (8.67) | -1.8 (8.41)

12. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 12
Description: Seventy-six joints were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score SJC of 0 (0 joints with swelling) to 76 (worst possible score/76 joints with swelling). Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 80
units on a scale | -3.6 (4.27) | -3.1 (5.64)

13. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 12
Description: The ASDAS is a continuous disease activity score: low score indicates lower disease activity and higher values indicate higher disease activity. The score ranges from 0 to no defined upper limit. It is categorized into 4 disease activity states based on score: inactive disease (< 1.3), moderate (≥ 1.3 to < 2.1), high (≥ 2.1 to ≤ 3.5), and very high (> 3.5). Clinically important and major improvements in ASDAS are defined as a reduction from Baseline of ≥ 1.1 and ≥ 2.0 points, respectively. Participants with non-missing Baseline and at least 1 non-missing post-Baseline value were included in post-Baseline visits. LOCF: missing value was imputed using the last non-missing post-Baseline value prior to missing value.
Time Frame: Baseline (last measurement prior to first DB dose), Week 12
Population: Efficacy analyses included all participants who were randomized and received at least 1 dose of double-blind study drug and with non-missing values for both Baseline and post-baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind (DB) Adalimumab | Double-blind Placebo
Number analyzed (Participants) | 84 | 80
units on a scale | -1.0 (1.07) | -0.5 (0.90)

ADVERSE EVENTS:
Time Frame: Baseline (day of first study drug administration) through Week 156 plus 70 days.
Groups:
- Double-blind Adalimumab: Adalimumab 40 mg subcutaneous (SC) injection every other week (eow) up to Week 12 in double-blind period.
- Any Adalimumab: All randomized participants who had received at least 1 dose of adalimumab (blinded or open-label) at any time during the study (up to Week 156).
Arm/Group | Double-blind Placebo | Double-blind Adalimumab | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/81 | 1/84 | 24/165
Other Adverse Events (participants affected / at risk) | 33/81 | 30/84 | 139/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=81) | Double-blind Adalimumab (N=84) | Any Adalimumab (N=165)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
ANAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 0 | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SPONDYLOARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PHAEOCHROMOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 0 | 1
VASCULITIS CEREBRAL (Nervous system disorders) | 0 | 0 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 0 | 1
RENAL DISORDER (Renal and urinary disorders) | 0 | 0 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=81) | Double-blind Adalimumab (N=84) | Any Adalimumab (N=165)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 4 | 12
DIARRHOEA (Gastrointestinal disorders) | 4 | 1 | 15
NAUSEA (Gastrointestinal disorders) | 3 | 2 | 10
FATIGUE (General disorders) | 1 | 1 | 14
BRONCHITIS (Infections and infestations) | 2 | 1 | 23
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 10
NASOPHARYNGITIS (Infections and infestations) | 11 | 4 | 51
PHARYNGITIS (Infections and infestations) | 0 | 0 | 12
RHINITIS (Infections and infestations) | 0 | 1 | 13
SINUSITIS (Infections and infestations) | 1 | 1 | 15
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 4 | 30
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 11
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 9
SPONDYLOARTHROPATHY (Musculoskeletal and connective tissue disorders) | 4 | 6 | 42
HEADACHE (Nervous system disorders) | 3 | 4 | 17
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 12
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 15
HYPERTENSION (Vascular disorders) | 0 | 2 | 12
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 7
INJECTION SITE REACTION (General disorders) | 0 | 1 | 8
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 6
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 8
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 6
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 8
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 6
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 6
DRY EYE (Eye disorders) | 1 | 1 | 5
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 6
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 5
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 7
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
CONJUNCTIVITIS (Infections and infestations) | 0 | 1 | 6
CYSTITIS (Infections and infestations) | 0 | 1 | 7
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 5
INFLUENZA (Infections and infestations) | 1 | 3 | 8
ORAL HERPES (Infections and infestations) | 0 | 1 | 5
TONSILLITIS (Infections and infestations) | 0 | 1 | 8
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.